CLINICAL TRIAL: NCT02989324
Title: Low Dose Vaginal Misoprostol With or Without Foley Catheter for Late Second Trimester Pregnancy Termination in Women With Previous Multiple Cesarean Sections
Brief Title: Vaginal Misoprostol and Foley Catheter for Late Second Trimester Termination of Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zuh- 4
Record Dates: First submitted 2016-11-30; First posted 2016-12-12 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2016-11

CONDITIONS: Late Second Trimester Termination of Pregnancy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Misoprosto (Experimental): Vaginal Misoprosto for Late Second Trimester Termination of Pregnancy With Previous Multiple Cesarean Section
  Interventions: Drug: MisoprostoL
- Misoprostol Plus Foley Catheter (Active Comparator): Misoprostol Plus Foley Catheter for Late Second Trimester Termination of Pregnancy With Previous Multiple Cesarean Sections
  Interventions: Drug: MisoprostoL; Device: Foley Catheter

INTERVENTIONS:
Drug: MisoprostoL — Vaginal MisoprostoL
  Other Names: CYTOTEC
Device: Foley Catheter — Misoprostol Plus Foley Catheter
  Arms: Misoprostol Plus Foley Catheter

SUMMARY:
Vaginal Misoprostol Versus Combined Low Dose Misoprostol Plus Foley Catheter for Late Second Trimester Termination of Pregnancy With Previous Multiple Cesarean Sections

DETAILED DESCRIPTION:
this study aims to compare between Vaginal Misoprostol and Combined Low Dose Misoprostol Plus Foley Catheter for Late Second Trimester Termination of Pregnancy With Previous Multiple Cesarean Sections to assess safety and efficacy of theses methods.

ELIGIBILITY:
Inclusion Criteria:late second trimester

* IUFD
* Previous Multiple Cesarean Sections

Exclusion Criteria:Low lying placenta

* asthma
* allergy to misoprostol
* patient refuse to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
induction to expulsion interval | 24 hours
  from time to start induction to time of complete expulsion of product of conception

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim A el sharkwy, MD, Principal Investigator — FACULTY OF MEDICINE ,ZAGAZIG UNIVERSITY
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No